CLINICAL TRIAL: NCT01117142
Title: A Study of the Kinetics of Lymphoid Cells in Patients With Monoclonal B-Cell Lymphocytosis (MBL), Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL), Mantle Cell Lymphoma (MCL) and Healthy Volunteers.
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Northwell Health (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100097; 10-H-0097
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Lymphoma, Mantle-cell; CLL (Chronic Lymphocytic Leukemia); Monoclonal B-Cell Lymphocytosis; Healthy Volunteers; Small Lymphocytic Lymphoma
Keywords: CLL (Chronic Lymphocytic Leukemia); Monoclonal B Cell Lymphocytosis; Small Lymphocytic Lymphoma; Mantle Cell Lymphoma; Cellular Proliferation; Chronic Lymphocytic Leukemia; CLL; Monoclonal B-Cell Lymphocytosis; MBL; SLL; MCL; Healthy Volunteer; HV
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Leukemia, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- CLL/SLL: Chronic lymphocytic leukemia/small lymphocytic lymphoma
- Healthy Volunteers: Healthy Volunteers
- MBL: Monoclonal B-cell lymphocytosis
- MCL: Mantle Cell Lymphoma

SUMMARY:
Background:

* Chronic lymphocytic leukemia (CLL), small lymphocytic lymphoma (SLL), and mantle cell lymphoma (MCL) are types of cancers in which there are too many abnormal lymphocytes (a type of white blood cell). Monoclonal B-cell lymphocytosis (MBL) is a condition in which the individual has a larger than normal number of lymphocytes. Individuals with CLL, SLL, MBL, and MCL may survive for many years without the need for treatment, but there is an apparent correlation between cell birth rates and disease activity. By studying the birth and death rates of lymphocytes, researchers hope to identify individuals who are at risk for worsening disease.
* Heavy water is similar in structure to regular water, but it has two deuterium atoms instead of two hydrogen atoms. Deuterium has one more neutron than hydrogen, which is what makes heavy water heavy. Heavy water is not radioactive, looks and tastes like regular water, and has no known harmful effects at research-level doses. When a small amount of heavy water is consumed daily, newly produced blood cells are labeled (tagged), which allows researchers to track cell growth and to measure the birth and death rates of CLL, SLL, MBL, MCL or normal lymphocytes.

Objectives:

- To study the birth and death rates of lymphocytes from individuals with MBL, CLL/SLL, and MCL, compared with lymphocytes from healthy volunteers.

Eligibility:

* Individuals at least 18 years of age who have been diagnosed with MBL, CLL, SLL, or MCL, but who have not been taking certain agents (Viagra, Levitra, Cialis, or other PDE-inhibitors, prednisone, cyclosporin-A, rapamycin, or other immunosuppressive agents, more than 2 cups of green tea daily, or Celebrex) for 4 weeks prior to enrollment in the study.
* Healthy volunteers at least 18 years of age, but who have not been taking certain agents (Viagra, Levitra, Cialis, or other PDE-inhibitors, prednisone, cyclosporin-A, rapamycin, or other immunosuppressive agents, more than 2 cups of green tea daily, or Celebrex)for 4 weeks prior to enrollment in the study.

Design:

* Participants will be screened with a medical history, physical examination, and initial blood tests. Other tests may be administered to the individuals with cancer, as required by the study researchers.
* All participants will drink regular doses of heavy water daily for a total of 4 weeks (labeling period). There is an optional 6-month follow-up or wash-out period during which no additional heavy water will be consumed.
* Blood samples will be collected weekly during the labeling period, and a bone marrow biopsy will be obtained where possible. Individuals with cancer may also have a lymph node biopsy during this part of the study.
* Additional blood samples may be collected during the optional wash-out phase of the study to determine the rate at which cancer cells disappear.
* Treatment is not provided as part of this protocol.

DETAILED DESCRIPTION:
Chronic lymphocytic leukemia (CLL) and its lymphoma variant, small lymphocytic lymphoma (SLL) were for decades considered diseases caused by the progressive accumulation of abnormal lymphocytes. The prevailing view being that CLL and SLL disease processes were driven by an underlying defect in apoptosis. While resistance to apoptosis appears to be important in the CLL and SLL disease process, recent studies suggest that cellular proliferation is more important than previously realized.

Cells from individuals with CLL who drank deuterated water (heavy water) for 6 weeks showed a turnover rate of 0.1 % to 1.1 % per day. In a second study involving CLL subjects who drank heavy water, average CLL turnover rates were in a similar range but approximately 2-fold lower than average B-cell turnover rates from healthy individuals. These studies have shown the safety and scientific value of using heavy water to study the kinetics of cell proliferation in patients and normal volunteers.

We now propose this study to expand on findings by other investigators. This study will address the site of proliferation for CLL/SLL cells and will include individuals with monoclonal B-cell lymphocytosis (MBL), a possible precursor of CLL. Furthermore, we will include patients with mantle cell lymphoma (MCL), a disease in which tumor proliferation plays an important role.

Study participants will drink heavy water daily for a total of 4 weeks (labeling period) with an optional 6 months follow up ( wash out period). Blood samples will be obtained weekly during the labeling period. A bone marrow and/or lymph node biopsy will be obtained where possible during the labeling period. Additional blood draws may be obtained during the optional wash-out phase of the study to determine the rate at which tumor cells disappear.

The primary objective of this exploratory study is to obtain an estimate of the proliferation rate of tumor cells in individuals with MBL, CLL/SLL, and MCL. Secondary objectives include the comparison of proliferation rates between different anatomic compartments, specifically peripheral blood, lymph node, and bone marrow and the estimation of the attrition or disappearance rate of cells during an optional phase of the protocol. Healthy volunteers may be included for comparison.

The primary objective of this exploratory study is to obtain an estimate of the proliferation rate of tumor cells in individuals with MBL, CLL/SLL, and MCL.

Secondary endpoints include: Proliferation rate in tissue compared to blood, disappearance rate of labeled cells from the blood and tissue, and the safety profile of heavy water in the study population.

ELIGIBILITY:
* INCLUSION CRITERIA: (MBL, CLL/SLL, MCL group)

4.1.1.<TAB>Diagnosed with MBL, CLL/SLL, or MCL

4.1.2.<TAB>Greater than or equal to 18 years of age

4.1.3.<TAB>Neutrophil count (ANC) greater than or equal to 1000/mcL

4.1.4.<TAB>Platelet count greater than or equal to 50K/mcL

EXCLUSION CRITERIA: (MBL, CLL/SLL, MCL group)

4.2.1.<TAB>Concomitant use of agents that have been described to affect the biology and/or proliferation rate of CLL cells but are not approved or accepted therapies for CLL, SLL, MCL, or MBL

* PDE-inhibitors (e.g. sildenafil, theophylline)
* Immunosuppressive agents (e.g., prednisone, cyclosporin-A, rapamycin)
* Green Tea extract (more than 2 cups per day)
* Cox-2 inhibitors

4.2.2.<TAB>Chronic or current clinically significant infection, including HIV or uncontrolled infection

4.2.3.<TAB>Receiving concurrent anticancer therapies

4.2.4.<TAB>Women who are pregnant or nursing, as well as women of childbearing potential who are unwilling to use a an agreed upon form of contraception for the duration of participation in this study

4.2.5<TAB>Sexually active males who are unwilling to follow the strict contraception requirements described in this protocol.

4.2.6<TAB>Inability to understand the investigational nature of the study, inability to provide informed consent

INCLUSION CRITERIA: (Healthy volunteer group)

4.3.1<TAB>Health status will be confirmed by brief History and Physical Exam and blood work

4.3.2<TAB>Greater than or equal to 18 years of age

4.3.3<TAB>CBC and coagulation panel within the expected normal ranges for the subject

EXCLUSION CRITERIA: (Healthy volunteer group)

4.4.1.<TAB>Concomitant use of agents that have been described to affect the biology and/or proliferation rate of CLL cells

* PDE-inhibitors (e.g. , slidenafil, theophylline)
* Immunosuppressive agents (e.g., cyclosporin-A, rapamycin)
* Green Tea extract (more than 2 cups per day)
* Cox-2 inhibitors

<TAB>

4.4.2.<TAB>Women who are pregnant or nursing, as well as women of childbearing potential who are unwilling to use an agreed upon form of contraception for the duration of study participation.

4.4.3<TAB> Sexually active males who are unwilling to follow the strict contraception requirements described in this protocol.

4.4.4.<TAB>Inability to understand the investigational nature of the study, inability to provide informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with eligible conditions or healthy volunteers aged 18 and over if participating as a normal volunteer who otherwise fulfill the eligibility criteria will be considered for the protocol.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-06-03 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the estimate of the cell proliferation rate of tumor cells in individuals with MBL, CLL/SLL, and MCL | 28 days
  Cell proliferation rate of tumor cells

SECONDARY OUTCOMES:
Secondary endpoints include: Proliferation rate in tissue compared to blood, disappearance rate of labeled cells from the blood and tissue and the safety profile of heavy water in the study population/ | 28 to 196 days

CONTACTS AND LOCATIONS:
Overall Officials: Clare C Sun, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hallek M, Bergsagel PL, Anderson KC. Multiple myeloma: increasing evidence for a multistep transformation process. Blood. 1998 Jan 1;91(1):3-21. PMID 9414264
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Thun MJ. Cancer statistics, 2009. CA Cancer J Clin. 2009 Jul-Aug;59(4):225-49. doi: 10.3322/caac.20006. Epub 2009 May 27. PMID 19474385
- [Background] Redaelli A, Laskin BL, Stephens JM, Botteman MF, Pashos CL. A systematic literature review of the clinical and epidemiological burden of acute lymphoblastic leukaemia (ALL). Eur J Cancer Care (Engl). 2005 Mar;14(1):53-62. doi: 10.1111/j.1365-2354.2005.00513.x. PMID 15698386
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2010-H-0097.html